CLINICAL TRIAL: NCT02229669
Title: Coronally Advanced Flap With Two Different Techniques for the Treatment of Multiple Gingival Recessions: A Split-mouth RCT
Brief Title: Coronally Advanced Flap With Two Different Techniques for the Treatment of Multiple Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Guilherme Barrella, MS, DDS, Paulista University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1158-9611
Record Dates: First submitted 2014-08-21; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Horizontal incisions (Experimental): Coronally advanced flap was performed by using horizontal interdental incisions. An initial horizontal incision was made slightly coronal to the CEJ from the distal to the mesial papilla of the teeth with the recessions. A second incision, 1 to 2 mm apart and parallel to the first incision, was made apically. A sulcular incision was made to link the second incisions and the blade was inserted extending beyond the mucogingival junction, to create a uniform split-thickness flap. The tissue between the two incisions was partially removed to obtain a uniform receptor site that permitted primary closure. Approximation sutures to place the edge of the flap at the base of the remaining papilla were performed.
  Interventions: Procedure: Horizontal incisions; Procedure: Oblique incisions
- Oblique incisions (Experimental): Coronally advanced flap was performed by using oblique incisions in interdental areas, according to the technique proposed by Zucchelli & De Sanctis (2000). Oblique submarginal interdental incisions were performed and continued with the intrasulcular incisions at the recession defects, resulting in a envelop flap that was raised with a split-full-split approach in the coronal-apical direction. During coronal advancement, each surgical papilla was dislocated with respect to the de-epithelized anatomic papilla by the oblique incisions. Interrupted sutures were performed to stabilize single surgical papilla over the interdental connective tissue bed.
  Interventions: Procedure: Horizontal incisions; Procedure: Oblique incisions

INTERVENTIONS:
Procedure: Horizontal incisions — Performed by using horizontal interdental incisions. An initial horizontal incision was made slightly coronal to the CEJ from the distal to the mesial papilla of the teeth with the recessions. A second incision, 1 to 2 mm apart and parallel to the first incision, was made apically. A sulcular incision was made to link the second incisions and the blade was inserted (2 to 3 mm) extending beyond the mucogingival junction (MGJ), to create a uniform split-thickness flap. The tissue between the two incisions was partially removed to obtain a uniform receptor site that permitted primary closure. Approximation sutures to place the edge of the flap at the base of the remaining papilla were performed. Passive closure of the wound margins without tension was achieved with interrupted coaptation.
Procedure: Oblique incisions — Coronally advanced flap was performed by using oblique incisions in interdental areas, according to the technique proposed by Zucchelli & De Sanctis (2000). Oblique submarginal interdental incisions were performed and continued with the intrasulcular incisions at the recession defects, resulting in a envelop flap that was raised with a split-full-split approach in the coronal-apical direction. During coronal advancement, each surgical papilla was dislocated with respect to the de-epithelized anatomic papilla by the oblique incisions. Interrupted sutures were performed to stabilize single surgical papilla over the interdental connective tissue bed.

SUMMARY:
This study compared the clinical outcomes of coronally advanced flap using two different surgical strategies in the treatment of multiple gingival recessions.

DETAILED DESCRIPTION:
The objective of this split-mouth, randomized controlled trial was to compare the clinical outcomes of coronally advanced flap (CAF) using two different surgical strategies in the treatment of multiple gingival recessions. Recessions were randomly treated according to a split-mouth design by means of: CAF with oblique interdental incisions (OBL technique) or CAF with horizontal interdental incisions (HOR technique). Marginal gingival recession (REC), clinical attachment level (CAL), pocket probing depth (PPD), height of keratinized tissue (HKT) and thickness of keratinized tissue (TKT) were measured at baseline, 3 and 6 months after treatment. Patient-centered outcomes concerning morbidity and improvement in the esthetic appearance were recorded using a Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy subjects
* Patients should have bilateral Class I and II MGRs (Miller 1985) in maxillary tooth (at least three recession-type defects affecting adjacent teeth in each side of the maxilla).
* At least 20 teeth and no sites with attachment loss and probing pocket depth (PPD) > 3 mm.
* Full-mouth plaque and bleeding on probing of < 20%.
* Involved tooth should present tooth vitality, absence of caries, restorations or extensive non-carious cervical lesion.

Exclusion Criteria:

* History of smoking.
* Antimicrobial and anti-inflammatory therapies in the previous 2 months.
* Previous mucogingival surgery at the region to be treated
* Systemic conditions that could affect tissue healing (e.g. diabetes).
* Use of orthodontic appliances.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Marginal gingival recession to 6 months | baseline, and at 3 and 6 months post-surgery

SECONDARY OUTCOMES:
height of keratinized tissue | Baseline, 3 and 6 months
thickness of keratinized tissue | baseline, 3 and 6 months
Clinical attachment level | baseline, 3 and 6 months
Probing deph | baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Suzana Pimentel, PHD, Principal Investigator — Paulista University; Guilherme Barrella, MS, Study Chair — Paulista University